CLINICAL TRIAL: NCT00238264
Title: A Phase II Study of Conformal Radiotherapy In Patients With Low-Grade Gliomas
Brief Title: Radiation Therapy in Treating Young Patients With Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0221; COG-ACNS0221 (Other: Clinical Trials.gov); CIRB-05016 (Other: Pediatric CIRB); CDR0000445095 (Other: Clinical Trials.gov)
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2016-11

CONDITIONS: Brain Tumor; Central Nervous System Tumor
Keywords: childhood oligodendroglioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; childhood low-grade cerebral astrocytoma; recurrent childhood visual pathway and hypothalamic glioma; untreated childhood cerebellar astrocytoma; untreated childhood visual pathway and hypothalamic glioma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Oligodendroglioma; Astrocytoma; Optic Nerve Glioma | interventions — Radiotherapy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (radiotherapy) (Experimental): Patients undergo reduced-field conformal radiation therapy 5 days a week for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy — Undergo 3D-CRT Undergo proton radiation therapy Undergo IMRT
  Other Names: 3-dimensional conformal radiation therapy; intensity-modulated radiation therapy; 3D conformal radiation therapy; 3D-CRT; IMRT

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase II trial is studying how well radiation therapy works in treating young patients with gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the marginal-failure rate in young patients with low-grade gliomas treated with reduced-field conformal radiotherapy.

Secondary

* Determine the progression-free survival, event-free survival, and overall survival rates of young patients treated with this regimen.
* Determine quality of life of patients treated with this regimen.
* Correlate MIB-1 labeling index with progression-free survival and overall survival of these patients.

OUTLINE: This is a multicenter study.

Patients undergo reduced-field conformal radiotherapy 5 days a week for 6 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline or 6 weeks after completion of study treatment and then at 2 and 5 years (closed as of 10/27/2010).

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* low-grade glioma, including any of the following:

  * Juvenile pilocytic astrocytoma (JPA) or pleomorphic JPA
  * Diffuse astrocytoma, including any of the following subtypes:

    * Fibrillary astrocytoma
    * Gemistocytic astrocytoma
    * Subependymal giant cell astrocytoma
    * Pleomorphic xanthoastrocytoma
  * Low-grade oligoastrocytoma
  * Low-grade oligodendroglioma
  * Low-grade glioma not otherwise specified NOTE: *Patients with chiasmatic lesions who have contiguous extension of tumor into other regions of the visual pathway by CT scan or MRI are eligible without histopathologic confirmation; repeat biopsy required for patients with recurrent tumors that enhance but whose initial tumor did not
* Measurable disease by radiography
* Meets any of the following criteria:

  * Progressive nonresectable disease

    * Any location in the brain
  * Patients with a less than gross total resection are eligible provided they are symptomatic from their tumor OR the risk from neurologic impairment with progression is high enough to warrant immediate treatment
  * Has undergone biopsy only
* Must have received ≥ 1 course of prior chemotherapy (for patients < 10 years of age)

  * Prior chemotherapy optional (for patients ≥ 10 years of age)
* No type-1 neurofibromatosis
* No evidence of leptomeningeal dissemination

PATIENT CHARACTERISTICS:

Age

* 3 to 20

Performance status

* ECOG 0-2 OR
* Karnofsky 50-100% (for patients > 16 years of age) OR
* Lansky 50-100% (for patients ≤ 16 years of age)

Life expectancy

* At least 1 year

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3 (transfusion independent)
* Hemoglobin ≥ 10.0 g/dL (transfusions allowed)

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* Not in status epilepticus, coma, or requiring assisted ventilation prior to study entry
* Patients with a seizure disorder are eligible provided they are on anticonvulsants AND disease is well controlled

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* Recovered from prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* Concurrent dexamethasone allowed provided patient has been on a stable dose for ≥ 2 weeks prior to study entry
* Concurrent dexamethasone allowed for symptoms of increased intracranial pressure

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics

Other

* No other concurrent anticancer therapy

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2006-11; Primary Completion 2013-12-30 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M. Cherlow, MD, Study Chair — Todd Cancer Institute at Long Beach Memorial Medical Center; Edward G. Shaw, MD, Study Chair — Wake Forest University Health Sciences
Locations (145):
- United States (127):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Keyser Family Cancer Center at Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Maimonides Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's - Dayton, Dayton, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Royal Children's Hospital, Brisbane, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (10):
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- New Zealand (3):
  - Starship Children's Health, Auckland
  - Christchurch Hospital, Christchurch
  - Wellington Children's Hospital, Wellington
- San Jorge Children's Hospital, Santurce, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Result] Ulin K, Urie MM, Cherlow JM. Results of a multi-institutional benchmark test for cranial CT/MR image registration. Int J Radiat Oncol Biol Phys. 2010 Aug 1;77(5):1584-9. doi: 10.1016/j.ijrobp.2009.10.017. Epub 2010 Apr 8. PMID 20381270

RESULTS

PARTICIPANT FLOW:
Groups:
- Reduced-field Conformal Radiation Therapy: Patients undergo reduced-field conformal radiation therapy 5 days a week for 6 weeks in the absence of disease progression or unacceptable toxicity.
  radiation therapy: Undergo 3D-CRT Undergo proton radiation therapy Undergo IMRT
Period: Overall Study
Arm/Group | Reduced-field Conformal Radiation Therapy
Started | 92
Completed | 56
Not Completed | 36
Not completed — Death | 7
Not completed — Lost to Follow-up | 18
Not completed — Withdrawal by Subject | 4
Not completed — Ineligible | 7

BASELINE CHARACTERISTICS:
Arm/Group | Reduced-field Conformal Radiation Therapy
Number analyzed (Participants) | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 86
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: Years] | 13.6 [4.4 to 20.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 82
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 75
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Marginal-failure Rate
Description: Patients who do not recur as well as those with either central or distant recurrence would be treatment successes for this endpoint. Monitoring will be based on a Bayesian rule, with binomial likelihood and a Beta on the parameter p, the proportion of failures that are marginal failures.
Time Frame: Up to 5 years
Population: All evaluable patients were included in this analysis (n = 84). One eligible patient was deemed to be not evaluable due to progression during treatment, and was excluded from the analysis per protocol.
Measure: Number; unit: percentage of failure rate
Groups:
- Reduced-field Conformal Radiation Therapy: Reduced-field conformal radiation therapy 5 days a week for 6 weeks
Arm/Group | Reduced-field Conformal Radiation Therapy
Number analyzed (Participants) | 84
percentage of failure rate | 0

2. Secondary Outcome: Progression-free Survival Probability
Description: To estimate the progression-free survival rate for patients with recurrent, progressive or symptomatic low-grade gliomas after treatment with reduced field conformal radiation.
Time Frame: 3 years
Population: All eligible patients were included in the analysis, per protocol.
Measure: Number (95% Confidence Interval); unit: Percentage 3-year PFS rate
Arm/Group | Reduced-field Conformal Radiation Therapy
Number analyzed (Participants) | 85
Percentage 3-year PFS rate | 77.1 [68.5 to 86.7]

3. Secondary Outcome: Event-free Survival Probability
Description: To estimate the event-free survival rate for patients with recurrent, progressive or symptomatic low-grade gliomas after treatment with reduced field conformal radiation
Time Frame: 3 years
Population: All eligible patients were included in the analysis, per protocol.
Measure: Number (95% Confidence Interval); unit: Percentage 3-year EFS rate
Arm/Group | Reduced-field Conformal Radiation Therapy
Number analyzed (Participants) | 85
Percentage 3-year EFS rate | 77.1 [68.5 to 86.7]

4. Secondary Outcome: Overall Survival Probability
Description: To estimate the overall survival rate for patients with recurrent, progressive or symptomatic low-grade gliomas after treatment with reduced field conformal radiation.
Time Frame: 3 years
Population: All eligible patients were included in the analysis, per protocol.
Measure: Number (95% Confidence Interval); unit: Percentage 3-year OS rate
Arm/Group | Reduced-field Conformal Radiation Therapy
Number analyzed (Participants) | 85
Percentage 3-year OS rate | 94.0 [89.1 to 99.2]

5. Secondary Outcome: Quality of Life (QOL)
Description: QOL accessed using the Behavior Assessment System for Children (BASC), the Adaptive Behavior Assessment System (ABAS), the Behavior Rating Inventory of Executive Function (BRIEF), and the Symptom Checklist-90-R (SCL-90-R).
Time Frame: Up to 5 years
Population: The QOL assessments were removed from the protocol as part of Amendment #1A (as of 10/27/2010) due to extremely low compliance. No QOL data were available for statistical analysis.
Arm/Group | Reduced-field Conformal Radiation Therapy
Number analyzed (Participants) | 0

6. Secondary Outcome: MIB-1 Labeling Index Using Immunohistochemical Techniques With the MIB-1 Antibody According to Established Methods
Description: The MIB-1 labeling Index will be calculated as the percentage of tumor nuclei that are immunoreactive.
Time Frame: At baseline
Population: All eligible patients with MIB-1 labeling index available.
Measure: Number (95% Confidence Interval); unit: percentage of tumor nuclei
Arm/Group | Reduced-field Conformal Radiation Therapy
Number analyzed (Participants) | 64
percentage of tumor nuclei | 3.1 [2.4 to 3.8]

7. Secondary Outcome: Correlation MIB-1 Labeling Index With PFS
Description: The primary methods of analysis will be via stratified Cox regression
Time Frame: Up to 10 years
Population: All eligible patients with MIB-1 data available were included in this analysis. Per protocol, patients were stratified by age and tumor location. Based on a predefined cutoff, patients were categorized as MIB high or low (high: >= 2; low: < 2). The hazard ratio below is for patients with MIB high (low is the reference level).
Measure: Number (95% Confidence Interval); unit: Hazard ratio
Arm/Group | Reduced-field Conformal Radiation Therapy
Number analyzed (Participants) | 64
Hazard ratio | 1.08 [0.42 to 2.81]

ADVERSE EVENTS:
Arm/Group | Reduced-field Conformal Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 5/85
Other Adverse Events (participants affected / at risk) | 5/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced-field Conformal Radiation Therapy (N=85)
Periorbital edema (Eye disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Abducens nerve disorder (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Oculomotor nerve disorder (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced-field Conformal Radiation Therapy (N=85)
Headache (Nervous system disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.